CLINICAL TRIAL: NCT06156306
Title: Effectiveness of CBT-I and CBT-I Combined ACT for Insomnia and Anxiety Symptoms in Youth: A Randomised Control Trial
Brief Title: CBT-I Versus CBT-I+ACT for Youths With Insomnia and Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN NGAN YIN, Assistant Professor, Department of Psychiatry, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230914
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Anxiety; Youth
Keywords: Insomnia; Anxiety; Youth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-I (Active Comparator): A total of 6 sessions of face-to-face group CBT-I therapy will be provided. Each session will last 90-120 mins, with each group 8-10 subjects.
  Interventions: Behavioral: CBT-I
- CBT-I combined ACT (Experimental): A total of 6 sessions of face-to-face group CBT-I+ACT therapy will be provided. Each session will last 90-120 mins, with each group 8-10 subjects.
  Interventions: Behavioral: CBT-I combined ACT

INTERVENTIONS:
Behavioral: CBT-I — The CBT-I intervention will cover sleep education, stimulus control, sleep restriction, cognitive therapy and relaxation training.
  Arms: CBT-I
Behavioral: CBT-I combined ACT — In addition to the standard CBT-I components, mindfulness, thought diary, and other ACT components will be taught in the group.
  Arms: CBT-I combined ACT

SUMMARY:
Insomnia in adolescents and youth is a long-standing public health concern due to its high prevalence and association with various physical and mental health problems. Insomnia and psychiatric disorders are highly comorbid and intercorrelated in adolescents. Among all mental disorders, anxiety has been shown to be have high comorbidity with insomnia, affecting approximately 30% of individuals. CBT for insomnia (CBT-I) has been shown to be effective in improving sleep complaints and short-term improvement in mood while previous systematic reviews of interventional studies have demonstrated the effectiveness of acceptance and commitment therapy (ACT) interventions in treating insomnia, both as a primary condition and with other physical and/or mental health comorbidities. This study aims to compare the effect of CBT-I and CBT-I combined ACT in improving anxiety symptoms in youth.

DETAILED DESCRIPTION:
Insomnia and psychiatric disorders are highly comorbid and intercorrelated in adolescents. Among all mental disorders, anxiety has been shown to be have high comorbidity with insomnia, affecting approximately 30% of individuals. Moreover, approximately three-quarters of anxious youth also report sleep-related problems. Literature reviews have investigated the relationship and the shared underlying mechanisms between sleep and anxiety. Anxiety sensitivity and pre-sleep arousal have been found to play a critical role in difficulty initiating sleep, which is the most common insomnia symptoms in adolescent population, partially due their natural delay of circadian rhythm. The findings suggest shared neurological and cognitive features that may account for dysregulation of both sleep and affect. Management targeting both sleep and anxiety is recommended due to potentially higher treatment efficacy and cost-effectiveness.

Accumulating evidence supports the effectiveness of cognitive-behavioural therapy for insomnia (CBT-I) and acceptance and commitment therapy (ACT) for addressing sleep and mood problems in adolescents. However, Only a few studies have directly compared the effectiveness of CBT-I and ACT. Past studies have shown that both CBT-I and ACT were effective in treating insomnia in adults.

This current study aims to compare the effect of CBT-I and CBT-I combined ACT in improving anxiety symptoms in youth. The primary hypothesis is that subjects in CBT-I combined ACT will have fewer anxiety symptoms as compared to CBT-I at post-intervention and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Youth who meet the following criteria would be eligible for taking part in this trial:

i. Chinese youth aged 15-24 years old, ii. Presence of insomnia problems as defined by insomnia severity index (ISI) using cut-off of 9, which has been locally validated cut off for detecting clinical insomnia), iii. Presence of anxiety features as defined by General Anxiety Disorder-7 (GAD-7) using cut-off of 10 for detecting clinical anxiety, iv. Ability to listen, speak, and read Chinese and Cantonese, and v. Written informed consent of participation into the study is given by youth and his/her parent's if under 18 years old; In addition, individual assent will also be obtained for subjects under age 18 years old vi. Possession of smartphone

Exclusion Criteria:

A youth would be excluded from the study if meeting one or more of the following criteria:

i. A clinical diagnosis of psychosis, schizophrenia, bipolar disorders, or intellectual disability ii. Having a diagnosed sleep disorder (e.g. delayed sleep phase and narcolepsy) that may potentially contribute to the disruption of sleep quantity and quality as determined by validated Diagnostic Interview for Sleep Patterns and Disorders (DISP) iii. Having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt) as assessed by The Structured Clinical Interview (SCID) iv. Currently receiving psychological treatment and/or pharmacological treatment for insomnia or anxiety disorder.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of anxiety symptoms and severity | Baseline, Postintervention (6 weeks), and 3-month follow up
  General Anxiety Disorder-7 (GAD-7) will be used to assess anxiety symptoms and severity.
Severity of anxiety symptoms | Baseline, Postintervention (6 weeks), and 3-month follow up
  Hospital Anxiety and Depression Scale (HADS) will be used to assess anxiety symptoms.
Clinician-rated severity of anxiety symptoms | Baseline, Postintervention (6 weeks), and 3-month follow up
  Hamilton Anxiety Rating Scale (HAM-A) will be used to assess anxiety symptoms.

SECONDARY OUTCOMES:
Severity of insomnia symptoms | Baseline, Postintervention (6 weeks), and 3-month follow up
  Insomnia Severity Index (ISI) will be used to measure the severity of insomnia symptoms.
Sleep-wake pattern | Baseline, Postintervention (6 weeks), and 3-month follow up
  Youths will be asked to keep a sleep diary to chart their daily sleep-wake pattern including sleep duration, wakeup time, bedtime and sleep latency
Daytime sleepiness | Baseline, Postintervention (6 weeks), and 3-month follow up
  Pediatric Daytime Sleepiness Scale (PDSS) will be used to assess adolescents' daytime sleepiness.
Anxiety trait | Baseline, Postintervention (6 weeks), and 3-month follow up
  The State-Trait Anxiety Inventory (STAI) will be used to measure anxiety trait
Severity of depressive symptoms | Baseline, Postintervention (6 weeks), and 3-month follow up
  Patient Health Questionnaire 9-item (PHQ-9) will be used to measure the severity of depressive symptoms.
Faulty sleep-related beliefs and cognitions | Baseline, Postintervention (6 weeks), and 3-month follow up
  Dysfunctional Beliefs and Attitudes about Sleep Scale-16-item (DBAS-16) will be used to measure faulty sleep-related beliefs and cognitions, which are cognitive aspects typically involved in the maintenance of insomnia.
Frequency of an individual practice sleep hygiene | Baseline, Postintervention (6 weeks), and 3-month follow up
  Sleep Hygiene Practice Scale (SHPS) will be used to measure the frequency of an individual practice sleep hygiene.
Psychological flexibility and experiential avoidance | Baseline, Postintervention (6 weeks), and 3-month follow up
  Acceptance and Action Questionnaire-II (AAQ-II) is related to the underlying ACT theory to measure psychological flexibility and experiential avoidance.
Individual's state of arousal | Baseline, Postintervention (6 weeks), and 3-month follow up
  Pre-Sleep Arousal Scale (PSAS) will be used to measure individual's state of arousal as one falls asleep.
Tendency to ruminate | Baseline, Postintervention (6 weeks), and 3-month follow up
  The Ruminative Responses Scale - short version (RRS-10) is a 10-item scale on a 4-likert scale. It measures the tendency to ruminate.
Major life events and hassles | Baseline, Postintervention (6 weeks), and 3-month follow up
  The Adolescent Stress Index (ASI), which was developed using a Hong Kong student sample, will be used to measure major life events and hassles
Global cognitive appraisal of one's life satisfaction | Baseline, Postintervention (6 weeks), and 3-month follow up
  The Satisfaction With Life Scale (SWLS): SWLS is a 5-item scale on a 7-Likert scale. It measures the global cognitive appraisal of one's life satisfaction.
Subjective well-being in the previous week | Baseline, Postintervention (6 weeks), and 3-month follow up
  The International Positive and Negative Affect Schedule Short Form (IPANAS-SF) will be used to capture the subjective well-being in the previous week. It has 9 items on a 5-Likert scale with previous study demonstrating satisfactory internal consistency reliability and reasonable nomological validity in Chinese youth.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Ngan Yin Chan, PhD, Principal Investigator — Department of Psychiatry, the Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, the Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No